CLINICAL TRIAL: NCT06523725
Title: A Randomized Controlled Trial Investigating the Safety and Efficacy of BRC-003 in Refractory Post-Traumatic Epilepsy
Brief Title: Trial Investigating the Safety and Efficacy of BRC-003 in Refractory Post-Traumatic Epilepsy
Acronym: PTE
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Company decision
Sponsor: Dr. Paul Lyons (Other)
Collaborators: Biopharmaceutical Research Company (Unknown)
Responsible Party: Sponsor-Investigator, Dr. Paul Lyons, Principal Investigator, Valley Health System
Organization: Valley Health System (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VHS-LY01
Record Dates: First submitted 2024-07-15; First posted 2024-07-26 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2024-07

CONDITIONS: Post-traumatic Epilepsy
MeSH Terms: conditions — Epilepsy, Post-Traumatic | interventions — nabiximols; Cannabinoids

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Part A and Part B (Experimental): Interventions:
  Drug: BRC-003 (High Cannabidiol Botanical Extract) 100 mg/mL
  Interventions: Drug: PO BRC-003 (High Cannabidiol Cannabis Extract)
- Part B (Placebo Comparator): Placebo Comparator: 1 Placebo Half of the patients will receive PO placebo
  Interventions:
  Drug: Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: PO BRC-003 (High Cannabidiol Cannabis Extract) — The research is divided into two phases: an open-label dose-finding phase (Part A) and a subsequent randomized controlled phase (Part B).
  Other Names: CBD, Cannabis Extract, Cannabinoids
  Arms: Part A and Part B
Drug: Placebo — Placebo
  Arms: Part B

SUMMARY:
This prospective double blind phase II study seeks to evaluate the safety and efficacy of BRC-003, a high CBD investigational product, in the treatment of refractory PTE (Post-Traumatic Epilepsy). The research is divided into two phases: an open-label dose-finding phase (Part A) and a subsequent randomized controlled phase (Part B). This design aims to provide a thorough understanding of the investigational product's impact on seizure frequency, seizure severity, mood, anxiety, sleep, and quality of life.

DETAILED DESCRIPTION:
Post-traumatic epilepsy (PTE) is a debilitating disorder characterized by recurrent seizures that develop following traumatic brain injury (TBI). Approximately 30 to 50% of patients with PTE may develop refractory epilepsy, wherein seizures persist despite treatment with multiple antiseizure medications (ASMs) or other therapeutic intervention. Moreover, the debilitating side effects of some ASMs can impact treatment compliance and patient quality of life; the side effects of ASMs may be more severe in patients with PTE.

Cannabis sativa L. has an extensive history of medical and therapeutic use. Growing interest in the utility of cannabinoids for medical indications including epilepsy, pain, nausea, appetite stimulation, muscle spasticity, and psychological disorders has led to its legalization in at least 14 countries as well as the regulatory approval of cannabis extract preparations, synthetic cannabinoids, and analogues. Cannabidiol (CBD), a non-intoxicating cannabinoid, has shown significant anticonvulsant properties and has received FDA (Food and Drug Administration) approval in three refractory seizure disorders.

This prospective study seeks to evaluate the safety and efficacy of BRC-003, a high CBD investigational product, in the treatment of refractory PTE. The research is divided into two phases: an open-label dose-finding phase (Part A) and a subsequent randomized controlled phase (Part B). This design aims to provide a thorough understanding of the investigational product's impact on seizure frequency, seizure severity, mood, anxiety, sleep, and quality of life.

ELIGIBILITY:
Inclusion Criteria:

Participants must meet all of the following criteria to be eligible for enrollment into the study:

1. Diagnosis consistent with PTE,

   - and -
2. History of a trial of at least two AEDs, including one trial of a combination of two concomitant AEDs, without successful seizure control. Vagus nerve stimulation (VNS), RNS, deep brain stimulation (DBS), or the ketogenic diet can be considered an equivalent to a drug trial,
3. Between 1-4 baseline anti-epileptic drugs at stable doses for a minimum of 4 weeks prior to enrollment,
4. VNS, DBS, or RNS must be on stable settings for a minimum of 3 months,
5. If on ketogenic diet, must be on stable ratio for a minimum of 3 months.
6. If applicable, documentation (including date of surgery) of prior VNS, DBS, RNS, Corpus Callosotomy, or other epilepsy surgery the patient has received.
7. Age 18 years and older
8. Acceptable method of contraception (or abstinence) for women of childbearing potential and for male patients with partners of childbearing potential; female patients must have a negative urine pregnancy test on the day of initiating IMP.
9. Weight ≥ 40 kg

Exclusion Criteria:

* Participants meeting any of the following criteria will not be eligible for participation in the study:

  1. Active psychogenic non-epileptic seizures (PNES),
  2. Patients who are pregnant, breastfeeding, or not using acceptable methods of contraception during the course of the study and for three months thereafter,
  3. Male patient's partner is of childbearing potential; unless willing to ensure that they (male patients) or their partner(s) are using acceptable methods of contraception during the course of the study and for three months thereafter,
  4. Use of medical marijuana, cannabis, hemp, or CBD based product in the previous 30 days, or during the study.
  5. Weight ≤ 40 kg
  6. Initiation of felbamate within the last 12 months,
  7. Allergy to CBD or any cannabis-type products,
  8. ALT >5 × ULN or AST >5 × ULN, as seen in participant's laboratory results,
  9. Hemoglobin <10 or hematocrit <30 or WBC < 2000, as seen in participant's laboratory results,
  10. Current (as assessed via C-SSRS) or history of suicidal ideation or attempt,
  11. In PI's judgment, active medical condition/treatment that impacts study activities,
  12. Unable to provide consent,
  13. No access to a mobile phone, and internet, not willing or able to download the eDiary application,
  14. Inability or failure to comply with study visits, requirements and/or instructions, and
  15. For Part B, prior enrollment in Part A of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-11-01 (Actual); Primary Completion 2025-04-15 (Actual); Study Completion 2025-04-15 (Actual)

PRIMARY OUTCOMES:
Safety assessment | Day 84
  Adverse events (AEs) and serious AEs (SAEs). The incidence of adverse events as measure of subject safety [Time Frame: Day 0 - Day 84] The number of subjects who experienced an adverse event during the study.
  * Vital signs
  * Laboratory assessments
Efficacy assessment | Day 84
  Change from baseline to 12 weeks (post-treatment) in number of Post-Traumatic Epilepsy (PTE) -associated seizures

SECONDARY OUTCOMES:
Number of patients considered treatment responders defined as those with a ≥ 50% reduction in PTE-associated seizure frequency. | Day 84
  Measured by the number of patients considered treatment responders
Number of patients considered treatment responders defined as those with a ≥ 25%, ≥ 50%, ≥ 75% or 100% reduction in PTE-associated seizure frequency. | Day 84
  Measured by the number of patients considered treatment responders
Number of patients experiencing a > 25% worsening, - 25 to + 25% no change, 25-50% improvement, 50-75% improvement or > 75% improvement in PTE-associated seizure frequency | Day 84
  Measured by the number of patients considered treatment responders
Change in number of PTE-associated seizure-free days. | Day 84
  per medical chart review
Seizure severity | Day 84
  via the Seizure Severity Questionnaire (SSQ). Minimum value: 11, Maximum value: 77. The lower the score, the better the outcome.
Emotional distress/depression Information System (PROMIS) Short Form | Day 84
  via the Patient-Reported Outcomes Measurement. Minimum score: 4, Maximum score: 20. The lower the score, the better the outcome.
Sleep disturbance | Day 84
  via the PROMIS Short Form. Minimum score: 4, Maximum score: 20. The lower the score, the better the outcome.
Performance of Social Roles and Activities | Day 84
  via the PROMIS Short Form. Minimum score: 4, Maximum score: 20. The lower the score, the better the outcome.
Anxiety | Day 84
  via the General Anxiety Disorder-7 (GAD-7) scale. 0-4: minimal anxiety, 5-9: mild anxiety, 10-14: moderate anxiety, 15-21: severe anxiety
Quality of life measurement | Day 84
  via QOLIE-31. Contains 17 multi-item measures of overall quality of life, emotional well-being, role limitations due to emotional problems, social support, social isolation, energy/fatigue, worry about seizure, medication effects, health discouragement, work/driving/social function, attention/concentration, language, memory, physical function, pain, role limitations due to physical problems, and health perceptions.
Use and effectiveness and of concomitant and frequency of rescue medications. | Day 84
  per medical chart review

CONTACTS AND LOCATIONS:
Overall Officials: Paul D Lyons, MD. PhD, Principal Investigator — Valley Health System
Locations (1):
- Winchester Medical Center, Winchester, Virginia, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] (Irimia & Van Horn, 2015; Wang et al., 2017)
- [Background] (Ding et al., 2016).